CLINICAL TRIAL: NCT02183701
Title: A Prospective Randomised Open-Label Blinded Endpoint Trial Comparing Telmisartan 80 mg and Losartan 50 mg + Hydrochlorothiazide 12.5 mg (Fixed Dose Combination) in Patients With Mild-to-Moderate Essential Hypertension Using Ambulatory Blood Pressure Monitoring
Brief Title: Telmisartan Compared to Losartan + Hydrochlorothiazide in Patients With Mild-to-moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.257
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; hydrochlorothiazide, losartan drug combination

ARMS (2):
- Telmisartan (Experimental): 4 weeks placebo run-in, 6-weeks fixed dose period
  Interventions: Drug: Telmisartan; Drug: Placebo
- Losartan + Hydrochlorothiazide (Active Comparator): 4 weeks placebo run-in, 6-weeks fixed dose period (Losartan 50 mg / HCTZ 12.5 mg)
  Interventions: Drug: Losartan + Hydrochlorothiazide; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Losartan + Hydrochlorothiazide
  Arms: Losartan + Hydrochlorothiazide
Drug: Placebo

SUMMARY:
The general aim and clinical objective of this trial is to determine the effect of telmisartan 80 mg compared to losartan 50 mg + HCTZ (Hydrochlorothiazide) 12.5 mg on reduction of blood pressure (BP) in patients with mild to moderate hypertension as assessed by 24 hour Ambulatory Blood Pressure Monitoring (ABPM) and trough sitting BP cuff measurements at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate essential hypertension defined as a mean seated diastolic blood pressure measurement of ≥ 95 mmHg measured by manual cuff sphygmomanometer, on Visit 2 of the four-week placebo run-in period (baseline)
* Mean seated systolic blood pressure ≥ 140 mmHg, measured by manual cuff at baseline (Visit 2)
* A 24-hour mean diastolic blood pressure , measured by ABPM, of ≥ 85 mmHg evaluated at baseline (Visit 3)
* Age 18 or older
* Patient's written informed consent in accordance with GCP (Good Clinical Practice) and local legislation

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to date of consent):

  * Who are not surgically sterile (hysterectomy, tubal ligation)
  * Who are NOT practising acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the trial. Acceptable methods of birth control include IUD (intrauterine device), oral, implantable or injectable contraceptives
  * Who have a positive urine pregnancy test
  * Who are nursing
* Mean seated diastolic blood pressure (DBP) > 114 mmHg or mean seated systolic BP > 200 mmHg, by manual cuff
* Any known hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * SGPT (serum glutamate pyruvate transaminase) (ALT) or SGOT (serum glutamate oxaloacetate transaminase) (AST) greater than two times the upper limit of normal
  * Serum creatinine > 1.8 mg/dl (or 159 µmol/l)
* Clinically relevant hypokalemia
* Known or suspected secondary hypertension
* Known bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney.
* Congestive heart failure (CHF) (NYHA (New York Heart Association) class CHF III-IV)
* Unstable angina within the past 3 months; stable angina where a change in nitrate therapy (dose or frequency) during the run-in period was required
* Stroke within the past 6 months prior to start of run-in period
* Myocardial infarction or cardiac surgery within the past 3 months prior to start of run-in period
* PTCA (percutaneous transluminal coronary angioplasty) within the past 3 months prior to start of run-in period
* Previous history of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
* Patients with unstable insulin-dependent diabetes mellitus (risk of hypoglycemia or HbA1c ≥ 10 % in history within 6 months prior to start of run-in period)
* Known drug or alcohol dependency within the past 6 months period prior to start of run-in period
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Patients receiving any investigational therapy within one month of signing the informed consent form
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of trial medication
* Concomitant use of lithium or cholestyramine or colestipol resins (potential drug interactions with HCTZ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 1998-04; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hour mean diastolic blood pressure measured by ABPM | Baseline (Day 28 of run-in period) and day 42

SECONDARY OUTCOMES:
Change from baseline in 24-hour mean systolic blood pressure measured by ABPM | Baseline (Day 28 of run-in period) and day 42
Change from baseline in systolic and diastolic blood pressures during other time periods during the 24-hour ABPM profile | Baseline (Day 28 of run-in period) and day 42
Change from baseline (Visit 2) in trough systolic and diastolic blood pressures measured by cuff sphygmomanometer | Baseline (Day 28 of run-in period) and day 42
Number of patient with of adverse events | up to 10 weeks
Changes from baseline in pulse rate | Baseline (Day 28 of run-in period) and day 42
Changes in physical examination | Screening and day 43
Changes in laboratory parameters | Screening and day 43
Changes in 12-lead electrocardiogram (ECG) | Baseline (Day 29 of run-in period) and day 43